CLINICAL TRIAL: NCT02662855
Title: Efficacy of Favipiravir Against Severe Ebola Virus Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Institute of Pharmacology and Toxicology (Other)
Collaborators: Beijing 302 Hospital (Other); 307 Hospital of PLA (Other); Sierra Leone-China Friendship Hospital (Unknown); Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPT-125
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Ebola Virus Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — favipiravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): WHO-recommended therapies, mainly symptomatic and supportive treatments. Briefly: body fluid management (intravenous or oral, depending on patient status), balanced nutrition (including glucose, electrolytes, vitamin, et al.), preventing intravascular volume depletion, correcting profound electrolyte abnormalities, avoiding the complications of shock, defervesce, anti-diarrheal, acesodyne, anti-anxiety. For patients with positive Plasmodium detection or bacterial infection, apply artemether-lumefantrine or antibiotics respectively. Details refer to 'Manual for the care and management of patients in Ebola Care Units/Community Care Centres, Interim emergency guidance' and 'Clinical Management of Patients with Viral Haemorrhagic Fever: A Pocket Guide for the Front-line Health Worker' by WHO.
  Interventions: Other: WHO-recommended therapies
- Treatment (Experimental): WHO-recommended therapies plus oral administration of Favipiravir
  Interventions: Other: WHO-recommended therapies; Drug: Favipiravir

INTERVENTIONS:
Other: WHO-recommended therapies — symptomatic and supportive treatments according to the WHO manual
Drug: Favipiravir — oral administration of Favipiravir tablets
  Other Names: T-705
  Arms: Treatment

SUMMARY:
The purpose of this study is to explore the therapeutic efficacy of Favipiravir, a broad-spectrum antiviral drug against severe cases of Ebola Virus Disease (EVD), which is the most difficult aspect for clinical management of EVD due to its high fatality rate.

DETAILED DESCRIPTION:
This is a prospective, open-label, controlled phase 2 trial of Favipiravir among severe cases (cases with hemorrhage, severe dehydration, consciousness disorders, shock, and high blood viral load with Ct value below 20) of confirmed EVD patients in the capital area of Sierra Leone. Patients with 13 years of age or older would be assigned in an 1:1 randomised manner to receive WHO-recommended therapy (mainly symptomatic and supportive therapies, control group. WHO, World Health Organization.) or oral Favipiravir (1600 mg twice on the first day, followed by a twice-daily dose of 600 mg until negative blood viral load detection or death) plus WHO-recommended therapy (treatment group). The primary efficacy end point was case fatality rate.The secondary efficacy endpoint is blood (plasma)viral load. Optimal inclusion number is 240 cases (120 for each group), but considering the actual situation of pandemic area, the front line doctors have the right to reset the inclusion number, and modify the study protocol according to the actual situation in the front.

ELIGIBILITY:
Inclusion Criteria:

* Male or famale，13 -75 years of age
* Clinical diagnosis of EVD
* Positive blood viral RNA detection
* With any one of the symptoms below:

Hemorrhage (including hematemesis, hemoptysis, hematochezia, hematuria, mucocutaneous hemorrhage), severe dehydration (including oliguria, anuria, feebleness, hypotension, tachycardia), consciousness disorders (including coma, delirium, confusion, convulsion), shock, and high blood viral load (Ct value below 20)

* Not received any therapies for EVD
* Provided written informed consent, by guardian or the patient himself
* Be able to administrate and tolerate oral administration of tablets

Exclusion Criteria:

* Severe vomiting
* Pregnancy and breast-feeding
* Received antiviral treatment against EVD

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Case fatality rate | 14 days

SECONDARY OUTCOMES:
Blood viral load | 1-3 days
  Described by Ct (cycle threshold) value

CONTACTS AND LOCATIONS:
Overall Officials: Wu Zhong, PhD, Principal Investigator — Beijing Institute of Pharmacology and Toxicology